CLINICAL TRIAL: NCT03203473
Title: Phase II Study of Optimized Management of NIVOlumab Based on REsponse in Patients With Advanced Renal Cell Carcinoma (OMNIVORE Study)
Brief Title: Study of Optimized Management of Nivolumab Based on Response in Patients With Advanced RCC (OMNIVORE Study)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Toni Choueiri, MD (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Toni Choueiri, MD, Sponsor Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-064
Record Dates: First submitted 2017-05-25; First posted 2017-06-29 (Actual); Results first posted 2022-04-25 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Renal Cancer
Keywords: Renal Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Overall cohort: Initial Primary Treatment with Nivolumab (induction phase) (Experimental): * Therapy with nivolumab IV every 2 weeks
  * Serial imaging assessments every 8 weeks
  * After confirmatory scans, patients are assigned to Arm A or Arm B.
  Interventions: Drug: Nivolumab
- Arm A: Observation Arm (for patients with persistent response to induction nivolumab) (Experimental): Patients with persistent response (complete or partial response) to induction nivolumab are assigned to Arm A (Observation Arm).
  * Patients discontinued nivolumab after allocation to Arm A.
  * Serial imaging assessments every 8 weeks.
  * If scans persistently show PR/CR, patients remained on observation.
  * If progressive disease develops, therapy with nivolumab (480 mg IV every 4 weeks) will be resumed.
  * If there is subsequent progression on nivolumab monotherapy, ipilimumab (1 mg/kg IV every 3 weeks x 2 doses) is added.
  * If progression after nivolumab + ipilimumab, therapy discontinued. If SD/PR/CR, nivolumab is continued until progression.
  Interventions: Drug: Ipilimumab; Drug: Nivolumab
- Arm B: Nivolumab+Ipilimumab then nivolumab alone (for patients with SD/PD to induction nivolumab) (Experimental): Patients with confirmed SD/PD to induction nivolumab are allocated to Arm B (Combination Therapy Arm).
  * In combination therapy, patients received nivolumab 3 mg/kg and ipilimumab 1 mg/kg intravenously every 3 weeks for two doses.
  * After then nivolumab will be continued at 480 mg IV every 4 weeks until disease progression.
  * Arm B patients undergo imaging at 12 weeks and then every 8 weeks.
  Interventions: Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Ipilimumab — YERVOY is thought to work with the body's immune system to increase the activity of T cells and cause the body to attack cancer cells
  Other Names: Yervoy
  Arms: Arm A: Observation Arm (for patients with persistent response to induction nivolumab); Arm B: Nivolumab+Ipilimumab then nivolumab alone (for patients with SD/PD to induction nivolumab)
Drug: Nivolumab — Nivolumab binds to and blocks the activation of PD-1, an Ig superfamily transmembrane protein, by its ligands programmed cell death ligand 1 (PD-L1), overexpressed on certain cancer cells, and programmed cell death ligand 2 (PD-L2), which is primarily expressed on APCs
  Other Names: Opdivo

SUMMARY:
This research study is studying two drugs at different time points as a possible treatment for advanced renal cell cancer

The drugs involved in this study are:

Nivolumab Ipilimumab

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of investigational drugs to learn whether the drugs work in treating a specific disease. "Investigational" means that the intervention is being studied.

Nivolumab and ipilimumab are antibodies (a type of human protein) that work to stimulate your body's immune system to fight tumor cells. The FDA (the U.S. Food and Drug Administration) has approved nivolumab as a treatment option for this disease; however, the FDA has not approved the way nivolumab and ipilimumab are being administered in this study. Ipilimumab is FDA approved for the treatment of melanoma (skin cancer) and has been previously studied in renal cell cancer.

This study is being done to evaluate nivolumab treatment strategies based on each patients individual response to treatment. In participants who have a response to treatment, nivolumab will be stopped and participants will be closely monitored. In participants who do not have a response to treatment,the investigators will investigate whether the addition of ipilimumab improves a participant response to treatment. Participant blood and tissue samples will be collected to learn about how certain biomarkers and genes relate to participant outcomes.

ELIGIBILITY:
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of ≤ 2 within 28 days prior to registration.
* Unresectable advanced or metastatic RCC to include both clear cell and non-clear histologies.

oPatients who have suspected metastatic RCC, which has not yet been pathologically proven, may be enrolled if they plan to undergo a cytoreductive nephrectomy, metastectomy, or biopsy. Fresh tissue from one of these procedures can be used for the clinical trial requirements (eligibility #4) as well as serve as pathologic confirmation of RCC. The pathologic confirmation must be documented prior to C1D1.

* Availability at the study site of formalin-fixed, paraffin-embedded (FFPE) archival tumor specimens, when available, and willingness of the subject to undergo mandatory fresh tumor biopsy prior to treatment initiation unless determined medically unsafe or not feasible. If a target lesion is biopsied at screening, this lesion must be followed as non-target lesion after the biopsy unless it is the patient's only target lesion. If there is only one target lesion, it should be followed as a target lesion regardless.

  * The archival specimen must contain adequate viable tumor tissue.
  * The specimen may consist of a tissue block (preferred and should contain the highest grade of tumor) or at least 30 unstained serial sections. Fine-needle aspiration, brushings, cell pellet from pleural effusion, bone marrow aspirate/biopsy are not acceptable.
* Previously untreated or treated subjects with no limit on prior lines of systemic therapies are allowed. Patient may have received prior adjuvant therapy.
* Measurable disease as defined by Response Evaluation Criteria In Solid Tumors RECIST 1.1 within 28 days prior to registration.

  * Demonstrate adequate organ function as defined in the table below. All screening labs to be obtained within 28 days prior to first study treatment.

System Laboratory Value

* Hematological

  * White blood cell (WBC) ≥ 2500 cells/µL
  * Absolute Neutrophil Count (ANC) ≥ 1500 cells/µL
  * Platelet count (plt) ≥ 100,000/ µL
  * Hemoglobin (Hgb) ≥ 9 g/dL (transfusions allowed)
  * Absolute lymphocyte count ≥ 500 cells/µL
* Renal

  --Serum creatinine OR Calculated creatinine clearance ≤ 1.5 x ULN ≥ 40 mL/min
* Cockcroft-Gault formula will be used to calculate creatinine clearance
* Hepatic and Other

  * Bilirubin ≤ 1.5 × upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) ≤ 2.5 × ULN
  * Alanine aminotransferase (ALT) ≤ 2.5 × ULN
  * Alkaline Phosphatase ≤ 2.5 × ULN
* Subjects with documented liver metastases should have AST and ALT ≤ 5 x ULN. Subjects with documented liver or bone metastases should have alkaline phosphatase ≤ 5 x ULN
* Subjects with known Gilbert's disease should have a serum bilirubin ≤ 3 x ULN.

  --Albumin > 2.5 g/dL
* Coagulation

  * International Normalized Ratio (INR) or Prothrombin Time (PT)
  * Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 × ULN (unless on prophylactic or therapeutic dosing with low molecular weight heparin)

    * Females of childbearing potential must have a negative serum pregnancy test within 28 days prior to registration. NOTE: Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.
    * Females of childbearing potential and males must be willing to abstain from heterosexual activity or to use 2 forms of effective methods of contraception from the time of informed consent until 120 days after treatment discontinuation. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method.
    * As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria

* Subjects meeting any of the criteria below may not participate in the study:
* Prior use of systemic checkpoint inhibitors for the management of metastatic RCC is excluded. Prior IFN-α or IL-2 is allowed.
* Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitors) within 2 weeks of enrollment or receipt of any anti-cancer therapy (including investigational therapy, monoclonal antibodies, cytokine therapy) within 4 weeks of enrollment.
* Treatment with systemic immunosuppressive medications including but not limited to:
* prednisone, dexamethasone, cyclosporin, azathioprine, methotrexate, thalidomide, anti- tumor necrosis factor (TNF) agents within 2 weeks of first study dose.
* Subjects who have received acute, low-dose systemic immunosuppressant medications may be enrolled (such as steroids for acute nausea or cancer-related pain ≤ 10 mg prednisone) may be enrolled sooner than 2 weeks of first study dose.
* Subjects with adrenal insufficiency on physiologic replacement doses of steroids may be enrolled (≤ 10 mg prednisone).
* The use of inhaled, topical, ocular or intra-articular corticosteroids and mineralocorticoids are allowed.
* Treatment with a receptor activator of nuclear factor kappa-B ligand (RANKL) inhibitor (e.g. denosumab) within 2 weeks of first study dose.
* Radiotherapy for RCC within 14 days of first study treatment with the exception of a single fraction of radiation administered for palliation of symptoms.
* Known active metastases to the brain, spinal cord or leptomeninges unless adequately treated with radiotherapy, radiosurgery, or surgery and stable for at least 4 weeks of first study treatment as documented by magnetic resonance imaging (MRI) or computerized tomography (CT) imaging and having no ongoing requirement for steroids.
* Malignancies other than RCC within 5 years of first study treatment with the exception of those with negligible risk of metastases or death and/or treated with expected curative outcome (carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer, ductal carcinoma in situ of the breast, non-muscle invasive urothelial carcinoma).
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion protein.
* Known hypersensitivity to any component of the nivolumab or ipilimumab product.
* Any active or recent history (within 6 months of first study dose) of autoimmune disease or syndrome that requires systemic corticosteroids (>10 mg daily prednisone equivalent) or immunosuppressive medications including but not limited to: myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with anti-phospholipid syndrome, Wegner's granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Subjects with vitiligo, controlled type I diabetes mellitus, hypo- or hyperthyroid disease, or surgical adrenal insufficiency requiring hormone replacement therapy are permitted to enroll.
* Any condition requiring treatment with corticosteroids (>10 mg daily prednisone equivalent) or other immunosuppressive medication within 14 days of the first dose of study drug. Inhaled, topical, ocular or intra-articular steroids and adrenal replacement steroid doses ≤ 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Uncontrolled adrenal insufficiency.
* History of idiopathic pulmonary fibrosis, organized pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening imaging CT of the chest. History of radiation pneumonitis in the radiation field is permitted.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome.
* Known active or chronic hepatitis B infection (defined as having a positive hepatitis B surface antigen (HBsAg) test at screening). Subject with past or resolved hepatitis B infection (defined as having a negative HBsAg test and positive antibody to hepatitis B core antigen test) are eligible. Hepatitis B viral DNA must be obtained in subjects with positive hepatitis B core antibody prior to first treatment start.
* Active hepatitis C infection. Subjects positive hepatitis C antibody test are eligible if PCR is negative for hepatitis C viral DNA.
* Severe infections within 4 weeks of first study treatment including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia.
* Receipt of therapeutic oral or IV antibiotics within 2 weeks of first study treatment. Subjects receiving routine antibiotic prophylaxis (for dental extractions/procedures) are eligible.
* Significant cardiovascular disease such as New York Heart Association (NYHA) class III or greater, myocardial infarction within the previous 3 months, unstable arrhythmias, unstable angina. Patients with known coronary artery disease, congestive heart failure not meeting the above criteria, or left ventricular ejection fraction < 45% must be on a stable regimen that is optimized in the opinion of the treating physician, in consultation with a cardiologist when appropriate.
* Prolonged corrected QT interval by the Fridericia correction formula (QTcF) on screening EKG > 500 msec.
* History of abdominal or tracheoesophageal fistula or GI perforation within 6 months of first study treatment.
* Clinical signs or symptoms of GI obstruction or requirement of routine parenteral nutrition.
* Evidence of abdominal free air not explained by paracentesis or recent surgical procedure.
* Serious, non-healing or dehiscing wound or active ulcer
* Major surgical procedure within 4 weeks of first study treatment.
* Presence of any toxicities attributed to prior anti-cancer therapy that are not resolved to grade 1 (National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0) or baseline before administration of study drug.
* Prior allogenic stem cell or solid organ transplant.
* Administration of a live, attenuated vaccine within 4 weeks for first study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2026-06-28 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Toni K Choueiri, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (8):
- United States (8):
  - University of California, San Diego Moores Cancer Center, La Jolla, California
  - University of Chicago Medical Center, Chicago, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Lifespan Comprehensve Cancer Center, Providence, Rhode Island
  - University of Utah, Huntsman Cancer Center, Salt Lake City, Utah
  - Unviersity of Wisconsin Carbone Cancer Center, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bootsma M, McKay RR, Emamekhoo H, Bade RM, Schehr JL, Mannino MC, Singh A, Wolfe SK, Schultz ZD, Sperger J, Xie W, Signoretti S, Kyriakopoulos CE, Kosoff D, Abel EJ, Helzer KT, Rydzewski N, Bakhtiar H, Shi Y, Blitzer G, Bassetti M, Floberg J, Yu M, Sethakorn N, Sharifi M, Harari PM, Choueiri TK, Lang JM, Zhao SG. Longitudinal Molecular Profiling of Circulating Tumor Cells in Metastatic Renal Cell Carcinoma. J Clin Oncol. 2022 Nov 1;40(31):3633-3641. doi: 10.1200/JCO.22.00219. Epub 2022 May 26. PMID 35617646
- [Derived] Bade RM, Schehr JL, Emamekhoo H, Gibbs BK, Rodems TS, Mannino MC, Desotelle JA, Heninger E, Stahlfeld CN, Sperger JM, Singh A, Wolfe SK, Niles DJ, Arafat W, Steinharter JA, Jason Abel E, Beebe DJ, Wei XX, McKay RR, Choueri TK, Lang JM. Development and initial clinical testing of a multiplexed circulating tumor cell assay in patients with clear cell renal cell carcinoma. Mol Oncol. 2021 Sep;15(9):2330-2344. doi: 10.1002/1878-0261.12931. Epub 2021 Mar 3. PMID 33604999
- [Derived] McKay RR, McGregor BA, Xie W, Braun DA, Wei X, Kyriakopoulos CE, Zakharia Y, Maughan BL, Rose TL, Stadler WM, McDermott DF, Harshman LC, Choueiri TK. Optimized Management of Nivolumab and Ipilimumab in Advanced Renal Cell Carcinoma: A Response-Based Phase II Study (OMNIVORE). J Clin Oncol. 2020 Dec 20;38(36):4240-4248. doi: 10.1200/JCO.20.02295. Epub 2020 Oct 27. PMID 33108238

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eighty-five patients were enrolled between October 2017 and July 2019 at 10 centers in the United States. Two patients never initiated treatment, resulting in 83 patients for analysis.
Groups:
- Overall Cohort: Initial Primary Treatment With Nivolumab (Induction Phase): * Therapy with nivolumab (480mg IV) every cycle (1cycle=4 weeks) up to 6 cycles
  * Serial imaging assessments every 8 weeks
  * After confirmatory scans, patients are assigned to Arm A or Arm B.
  Nivolumab: Nivolumab binds to and blocks the activation of PD-1, an Ig superfamily transmembrane protein, by its ligands programmed cell death ligand 1 (PD-L1), overexpressed on certain cancer cells, and programmed cell death ligand 2 (PD-L2), which is primarily expressed on APCs
- Arm A: Observation Arm (for Patients With Persistent Response to Induction Nivolumab): Patients with persistent response (complete or partial response) to induction nivolumab were assigned to Arm A (Observation Arm)
  * Serial imaging assessments every 8 weeks
  * If progressive disease develops, salvage therapy with nivolumab (480 mg IV every 4 weeks) will be resumed.
  * If there is subsequent progression on nivolumab monotherapy, ipilimumab (1 mg/kg IV every 3 weeks x 2 doses) is added.
  * If progression after nivolumab + ipilimumab, therapy discontinued. If SD/PR/CR, nivolumab is continued until progression.
- Arm B: Nivolumab+Ipilimumab Then Nivolumab Alone (for Patients With SD/PD to Induction Nivolumab): Patients with confirmed SD/PD to induction nivolumab were allocated to Arm B (Combination Therapy Arm).
  * In combination therapy, patients received nivolumab 3 mg/kg and ipilimumab 1 mg/kg intravenously every 3 weeks for two doses.
  * After then nivolumab will be continued at 480 mg IV every 4 weeks until disease progression.
  * Arm B patients underwent imaging at 12 weeks and then every 8 weeks.
Period: Induction phase
Arm/Group | Overall Cohort: Initial Primary Treatment With Nivolumab (Induction Phase) | Arm A: Observation Arm (for Patients With Persistent Response to Induction Nivolumab) | Arm B: Nivolumab+Ipilimumab Then Nivolumab Alone (for Patients With SD/PD to Induction Nivolumab)
Started | 85 | 0 | 0
Completed | 69 | 0 | 0
Not Completed | 16 | 0 | 0
Not completed — Never started primary treatment | 2 | 0 | 0
Not completed — Withdrew from study due to progressive disease | 7 | 0 | 0
Not completed — Withdrew from study due to toxicity | 7 | 0 | 0
Period: Arm Allocation Phase
Arm/Group | Overall Cohort: Initial Primary Treatment With Nivolumab (Induction Phase) | Arm A: Observation Arm (for Patients With Persistent Response to Induction Nivolumab) | Arm B: Nivolumab+Ipilimumab Then Nivolumab Alone (for Patients With SD/PD to Induction Nivolumab)
Started (All 85 patients were off primary treatment (induction phase), of whom, 69 patients entered the 2nd period (12 were allocated to Arm A and 57 were allocated to Arm B).) | 0 | 12 | 57
Completed | 0 | 0 | 0
Not Completed | 0 | 12 | 57
Not completed — Still on Arm A-observation | 0 | 7 | 0
Not completed — started salvage therapy | 0 | 5 | 0
Not completed — Disease progression | 0 | 0 | 37
Not completed — Adverse Event | 0 | 0 | 11
Not completed — Physician Decision | 0 | 0 | 3
Not completed — Death | 0 | 0 | 1
Not completed — Developed 2nd cancer | 0 | 0 | 1
Not completed — Intercurrent illness | 0 | 0 | 1
Not completed — Still on arm-B treatment | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Out of 85 patients enrolled, 83 patients received protocol treatment and were included for analysis; 2 patients who did not proceed with treatment were excluded from all analysis.
Groups:
- Overall Cohort: Initial Primary Treatment With Nivolumab (Induction Phase): * Therapy with nivolumab (480mg IV) every cycle (1cycle=4 weeks)
  * Serial imaging assessments every 8 weeks
  * After confirmatory scans, patients are assigned to Arm A or Arm B.
  Nivolumab: Nivolumab binds to and blocks the activation of PD-1, an Ig superfamily transmembrane protein, by its ligands programmed cell death ligand 1 (PD-L1), overexpressed on certain cancer cells, and programmed cell death ligand 2 (PD-L2), which is primarily expressed on APCs
Arm/Group | Overall Cohort: Initial Primary Treatment With Nivolumab (Induction Phase)
Number analyzed (Participants) | 83
Age, Continuous [Median (Full Range); unit: years] | 61 [33 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 75
  More than one race | 4
  Unknown or Not Reported | 1
Histology [Count of Participants; unit: Participants]
  Clear Cell | 80
  Non-clear Cell | 3
Previous systemic therapy [Count of Participants; unit: Participants]
  No | 42
  Yes | 41

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Persistent Partial Response (PR) or Complete Response (CR) at 1 Year Since Nivolumab Discontinuation (Arm A Only)
Description: Persistent PR or CR is defined per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 guidelines. Radiologic disease assessment was performed every 8 weeks after patients discontinued nivolumab induction therapy. At 1 year after nivolumab discontinuation, the percentage of patients with persistent PR and CR were reported (for Arm A only).
Time Frame: From nivolumab discontinuation until 1 year after discontinuation with nivolumab
Population: 12 patients were assigned to arm A after nivolumab induction therapy.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Arm A-Observation Arm (for Patients With Persistent Response to Induction Nivolumab): Patients with persistent response (complete or partial response) to induction nivolumab were assigned to Arm A (Observation Arm)
  * Serial imaging assessments every 8 weeks
  * If progressive disease develops, therapy with nivolumab (480 mg IV every 4 weeks) will be resumed.
  * If there is subsequent progression on nivolumab monotherapy, ipilimumab (1 mg/kg IV every 3 weeks x 2 doses) is added.
  * If progression after nivolumab + ipilimumab, therapy discontinued. If SD/PR/CR, nivolumab is continued until progression.
Arm/Group | Arm A-Observation Arm (for Patients With Persistent Response to Induction Nivolumab)
Number analyzed (Participants) | 12
percentage of participants | 42 [18 to 68]

2. Primary Outcome: Percentage of Subjects With Stable or Progressive Disease (SD/PD) to Nivolumab Induction That Convert to Complete or Partial Response (CR/PR) Upon the Addition of Ipilimumab to Nivolumab (Arm B Only)
Description: Response is defined per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 guideline. After initiation of ipilimumab, Arm B patients underwent imaging after the first 12 weeks and then every 8 weeks until disease progression. Best overall response during Arm B treatment were summarized with 90% confidence interval.
Time Frame: For arm B patients, from arm B treatment (nivolumab+ipilimumab) initiation until last imaging assessment during the treatment; assessed up to 22 months.
Population: 57 patients were assigned to Arm B after nivolumab induction therapy
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Arm B Nivolumab+Ipilimumab Then Nivolumab Alone (for Patients With SD/PD to Induction Nivolumab): Patients with confirmed SD/PD to induction nivolumab were allocated to Arm B (Combination Therapy Arm).
  * In combination therapy, patients received nivolumab 3 mg/kg and ipilimumab 1 mg/kg intravenously every 3 weeks for two doses.
  * After then nivolumab will be continued at 480 mg IV every 4 weeks until disease progression.
  * Arm B patients underwent imaging after the first 12 weeks and then every 8 weeks..
Arm/Group | Arm B Nivolumab+Ipilimumab Then Nivolumab Alone (for Patients With SD/PD to Induction Nivolumab)
Number analyzed (Participants) | 57
percentage of participants | 4 [1 to 11]

3. Secondary Outcome: Median Progression Free Survival (Arm B)
Description: Progression-free survival (PFS) for Arm B was defined as time from the start of arm B treatment until progression (by RECIST 1.1 or clinical PD) or death from any cause or censored at date of last disease evaluation for those who are alive and have not progressed. PFS distribution was estimated using the product-limit method of Kaplan-Meier, median and 95% confidence interval was reported.
Time Frame: After initiation of Arm B treatment, patients underwent imaging at 12 weeks and then every 8 weeks, up to 22 months.
Population: 57 patients were allocated to Arm B treatment after completing nivolumab induction
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm B Nivolumab+Ipilimumab Then Nivolumab Alone (for Patients With SD/PD to Induction Nivolumab)
Number analyzed (Participants) | 57
months | 4.7 [2.7 to 8.3]

4. Secondary Outcome: 18-month Overall Survival Rate From Initiation of Nivolumab Induction (Overall Cohort)
Description: Overall survival (OS) was defined as the time from initiation of nivolumab induction until death due to any cause or censored at date of last follow-up for surviving patients. OS rate was estimated using the product-limit method of Kaplan-Meier;18-month OS rate and 95% confidence interval were reported.
Time Frame: Patients were followed from initiation of Nivolumab induction until to death or date last known alive. Kaplan-Meier curve for OS assessed up to 28 months; the 18-month time point estimate for OS was reported.
Population: Out of 85 patients enrolled, 83 patients received nivolumab induction treatment and were included for analysis; 2 patients who did not proceed with treatment were excluded from all analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Initial Primary Treatment With Nivolumab (Induction Phase): * Therapy with nivolumab (480mg IV) every cycle (1cycle=4 weeks)
  * Serial imaging assessments every 8 weeks
  * After confirmatory scans, patients are assigned to Arm A or Arm B.
  Nivolumab: Nivolumab binds to and blocks the activation of PD-1, an Ig superfamily transmembrane protein, by its ligands programmed cell death ligand 1 (PD-L1), overexpressed on certain cancer cells, and programmed cell death ligand 2 (PD-L2), which is primarily expressed on APCs
Arm/Group | Initial Primary Treatment With Nivolumab (Induction Phase)
Number analyzed (Participants) | 83
percentage of participants | 79 [67 to 87]

5. Secondary Outcome: Percent of Subjects Who Were Free of Nivolumab Salvage Therapy at 1 Year Since Discontinuation of Nivolumab Induction (Arm A)
Description: Number and proportion of arm A patients who remained free of nivolumab treatment at 1 year since discontinuation of nivolumab induction
Time Frame: For arm A, from nivolumab discontinuation until 1 year after discontinuation with nivolumab
Population: 12 patients were allocated to arm A (observation arm) after nivolumab induction therapy.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A-Observation Arm (for Patients With Persistent Response to Induction Nivolumab)
Number analyzed (Participants) | 12
percentage of participants | 42 [18 to 68]

6. Secondary Outcome: Immune Related Objective Response Rate (irORR) in Arm A and Arm B
Description: The irORR is assessed according to immune-related Response Criteria (irRC).
  * Immune-Related Complete Response (irCR): Complete disappearance of all tumor lesions (index and non-index together with no new measurable/unmeasurable lesions) for at least 4 weeks from the date of documentation of complete response
  * Decrease, relative to baseline, of 50% or greater in the sum of the products of the two largest perpendicular diameters (SPD) of all target and all new measurable lesions in two consecutive observations not less than 4 weeks apart.
Time Frame: For arm A, radiology imaging will be done every 8 weeks until disease progression. For arm B, radiology imaging will be done at 12 weeks and then every 8 weeks until disease progression
Population: Since the trial was designed in 2015, immune-related response has been infrequently used in VEGF/IO trials for kidney cancer. Most RCC trials have mainly focused on the traditional RECIST-based response as the primary endpoint. Therefore, the study team did not pursue immune-related response assessment and that data was not collected.
Groups:
- Arm B- Nivolumab+Ipilimumab Then Nivolumab Alone (for Patients With SD/PD to Nivolumab Induction): Patients with confirmed SD/PD to induction nivolumab were allocated to Arm B (Combination Therapy Arm).
  * In combination therapy, patients received nivolumab 3 mg/kg and ipilimumab 1 mg/kg intravenously every 3 weeks for two doses.
  * After then nivolumab will be continued at 480 mg IV every 4 weeks until disease progression.
  * Arm B patients underwent imaging after the first 12 weeks and then every 8 weeks..
Arm/Group | Arm A-Observation Arm (for Patients With Persistent Response to Induction Nivolumab) | Arm B- Nivolumab+Ipilimumab Then Nivolumab Alone (for Patients With SD/PD to Nivolumab Induction)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percentage of Subjects Who Experience Grade 3-4 Treatment-related Adverse Event (TRAE) During the Nivolumab Induction Therapy (Overall Cohort)
Description: Adverse event was assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 4.
  The following AE attribution was considered as treatment-related:
  * Definite - The AE is clearly related to the study treatment.
  * Probable - The AE is likely related to the study treatment.
  * Possible - The AE may be related to the study treatment.
Time Frame: Adverse events during the nivolumab induction were measured from nivolumab initiation until 3 months following the last dose of nivolumab induction or until start of arm B treatment, assessed up to 9 months from nivolumab start
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Initial Primary Treatment With Nivolumab (Induction Phase): * Therapy with nivolumab (480mg IV) every cycle (1cycle=4 weeks) up to 6 cycles.
  * Serial imaging assessments every 8 weeks
  * After confirmatory scans, patients are assigned to Arm A or Arm B.
  Nivolumab: Nivolumab binds to and blocks the activation of PD-1, an Ig superfamily transmembrane protein, by its ligands programmed cell death ligand 1 (PD-L1), overexpressed on certain cancer cells, and programmed cell death ligand 2 (PD-L2), which is primarily expressed on APCs
Arm/Group | Initial Primary Treatment With Nivolumab (Induction Phase)
Number analyzed (Participants) | 83
percentage of participants | 7 [3 to 15]

8. Secondary Outcome: Percentage of Subjects Who Experienced Grade 3-4 Treatment Related Adverse Events (TRAE) During the Arm B Treatment (Arm B Only)
Description: as for outcome 7
Time Frame: For arm B, adverse events were measured from arm B treatment initiation until 3 months following the last dose of arm B treatment, assessed up to 26 months from arm B start
Population: 57 patients had been allocated to arm B after nivolumab induction therapy
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Arm B Nivolumab+Ipilimumab Then Nivolumab Alone (for Patients With SD/PD to Induction Nivolumab): Patients with confirmed SD/PD to induction nivolumab were allocated to Arm B (Combination Therapy Arm).
  * In combination therapy, patients received nivolumab 3 mg/kg and ipilimumab 1 mg/kg intravenously every 3 weeks for two doses.
  * After then nivolumab will be continued at 480 mg IV every 4 weeks until disease progression.
  * Arm B patients underwent imaging at 12 weeks and then every 8 weeks until disease progression.
Arm/Group | Arm B Nivolumab+Ipilimumab Then Nivolumab Alone (for Patients With SD/PD to Induction Nivolumab)
Number analyzed (Participants) | 57
percentage of participants | 25 [14 to 38]

9. Secondary Outcome: Percentage of Subjects Who Had Complete or Partial Response (CR/PR) to Nivolumab Induction Therapy According to International mRCC Database Consortium (IMDC) Risk Groups.
Description: Response (PR or CR) is defined per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1 guidelines. Radiologic disease assessment was performed every 8 weeks during the induction therapy with nivolumab.
Time Frame: From start of nivolumab induction until the discontinuation of nivolumab induction, assessed up to 7 months
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Initial Primary Treatment With Nivolumab (Induction Phase)
Number analyzed (Participants) | 83
percentage of participants
  IMDC favorable risk: number analyzed (Participants) | 27
  IMDC favorable risk | 11 [3 to 26]
  IMDC intermediate risk: number analyzed (Participants) | 45
  IMDC intermediate risk | 13 [6 to 25]
  IMDC poor risk: number analyzed (Participants) | 11
  IMDC poor risk | 9 [1 to 36]

10. Secondary Outcome: Percentage of Subjects Who Had Complete or Partial Response (CR/PR) to Nivolumab Induction Therapy According to Prior Treatment
Description: as for outcome 9
Time Frame: From start of nivolumab induction until the discontinuation of nivolumab induction, assessed up to 7 months
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Initial Primary Treatment With Nivolumab (Induction Phase)
Number analyzed (Participants) | 83
percentage of participants
  Treatment Naive: number analyzed (Participants) | 42
  Treatment Naive | 12 [5 to 23]
  Previously treated: number analyzed (Participants) | 41
  Previously treated | 12 [5 to 24]

11. Secondary Outcome: Percentage of Subjects Who Had Complete or Partial Response (CR/PR) to Nivolumab Induction Therapy According to Histology Type
Description: as for outcome 9
Time Frame: From start of nivolumab induction until the discontinuation of nivolumab induction, assessed up to 7 months
Population: Given the majority (96%) of patients had clear cell histology, subgroup analysis of response by histology type was not performed.
Arm/Group | Initial Primary Treatment With Nivolumab (Induction Phase)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Overall cohort (nivolumab induction): adverse event (AE) was measured from nivolumab start until 3 months following the last dose of nivolumab or until start of arm B treatment, up to 9 months from nivolumab start. Arm B (nivolumab+ipilimamab then nivolumab alone): AE was measured from arm B treatment start until 3 months following the last dose of arm B treatment, up to 26 months from arm B start. Arm A (observation arm): AE was not reported as patents were in observation arm.
Description: Overall cohort included 83 patients who received nivolumab, excluding 2 patients who did not receive treatment.
  Arm B: 57 patients on arm B were assessed for AE. Serious AEs included those with a severity grade of 3 or higher and a treatment attribution of possible, probable, or definite.
  Arm A:12 patients on arm A. AE was not reported since this was an observation arm. If a patient resumes therapy after progression to arm A, AE from subsequent therapy was not counted as arm A toxicities.
Groups:
- Overall Cohort: Initial Primary Treatment With Nivolumab (Induction Phase): * Therapy with nivolumab (480mg IV) every cycle (1cycle=4 weeks) up to 6 cycles.
  * Serial imaging assessments every 8 weeks
  * After confirmatory scans, patients are assigned to Arm A or Arm B.
  Nivolumab: Nivolumab binds to and blocks the activation of PD-1, an Ig superfamily transmembrane protein, by its ligands programmed cell death ligand 1 (PD-L1), overexpressed on certain cancer cells, and programmed cell death ligand 2 (PD-L2), which is primarily expressed on APCs
- Arm B: Nivolumab+Ipilimumab Then Nivolumab Alone (for Patients With SD/PD to Induction Nivolumab): Patients with confirmed SD/PD to induction nivolumab were allocated to Arm B (Combination Therapy Arm).
  * In combination therapy, patients received nivolumab 3 mg/kg and ipilimumab 1 mg/kg intravenously every 3 weeks for two doses.
  * After then nivolumab will be continued at 480 mg IV every 4 weeks until disease progression.
  * Arm B patients underwent imaging after the first 12 weeks and then every 8 weeks..
  Ipilimumab: YERVOY is thought to work with the body's immune system to increase the activity of T cells and cause the body to attack cancer cells
  Nivolumab: Nivolumab binds to and blocks the activation of PD-1, an Ig superfamily transmembrane protein, by its ligands programmed cell death ligand 1 (PD-L1), overexpressed on certain cancer cells, and programmed cell death ligand 2 (PD-L2), which is primarily expressed on APCs
- Arm A: Arm A-Observation Arm (for Patients With Persistent Response to Induction Nivolumab): Patients with persistent response (complete or partial response) to induction nivolumab are assigned to Arm A (Observation Arm).
  - AE was not reported since this was an observation arm. If a patient resumes nivolumab therapy after progression to arm A, AE from the subsequent therapy was not counted as arm A toxicities.
Arm/Group | Overall Cohort: Initial Primary Treatment With Nivolumab (Induction Phase) | Arm B: Nivolumab+Ipilimumab Then Nivolumab Alone (for Patients With SD/PD to Induction Nivolumab) | Arm A: Arm A-Observation Arm (for Patients With Persistent Response to Induction Nivolumab)
All-Cause Mortality (participants affected / at risk) | 19/83 | 12/57 | 1/12
Serious Adverse Events (participants affected / at risk) | 6/83 | 14/57 | 0/12
Other Adverse Events (participants affected / at risk) | 80/83 | 55/57 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Cohort: Initial Primary Treatment With Nivolumab (Induction Phase) (N=83) | Arm B: Nivolumab+Ipilimumab Then Nivolumab Alone (for Patients With SD/PD to Induction Nivolumab) (N=57) | Arm A: Arm A-Observation Arm (for Patients With Persistent Response to Induction Nivolumab) (N=12)
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Alkaline phosphatase increased (Investigations) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 2 | 0
CPK increased (Investigations) | 1 | 0 | 0
Creatinine increased (Investigations) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Eye disorders - Other, specify (Eye disorders) | 1 | 0 | 0
General disorders and administration site conditions - Other, specify (General disorders and administration site conditions) | 0 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 4 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Infusion related reaction (General disorders and administration site conditions) | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Portal hypertension (Hepatobiliary disorders) | 0 | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 1 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Cohort: Initial Primary Treatment With Nivolumab (Induction Phase) (N=83) | Arm B: Nivolumab+Ipilimumab Then Nivolumab Alone (for Patients With SD/PD to Induction Nivolumab) (N=57) | Arm A: Arm A-Observation Arm (for Patients With Persistent Response to Induction Nivolumab) (N=12)
Abdominal pain (Gastrointestinal disorders) | 4 | 3 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 3 | 0
Alanine aminotransferase increased (Investigations) | 9 | 6 | 0
Alkaline phosphatase increased (Investigations) | 4 | 2 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 11 | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 7 | 7 | 0
Anxiety (Psychiatric disorders) | 2 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 11 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 8 | 6 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 3 | 0
Bloating (Gastrointestinal disorders) | 3 | 1 | 0
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 2 | 0
Blood bilirubin increased (Investigations) | 3 | 0 | 0
Blurred vision (Eye disorders) | 1 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Bronchial infection (Infections and infestations) | 2 | 1 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0 | 0
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
CD4 lymphocytes decreased (Investigations) | 1 | 0 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Chills (General disorders and administration site conditions) | 1 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 3 | 0
Confusion (Psychiatric disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 7 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 9 | 0
Creatinine increased (Investigations) | 5 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 2 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 16 | 10 | 0
Dizziness (Nervous system disorders) | 2 | 3 | 0
Dry eye (Eye disorders) | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 5 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 | 2 | 0
Edema face (General disorders and administration site conditions) | 1 | 1 | 0
Edema limbs (General disorders and administration site conditions) | 6 | 2 | 0
Edema trunk (General disorders and administration site conditions) | 1 | 0 | 0
Endocrine disorders - Other, specify (Endocrine disorders) | 2 | 2 | 0
Eye disorders - Other, specify (Eye disorders) | 3 | 1 | 0
Facial muscle weakness (Nervous system disorders) | 1 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fatigue (General disorders and administration site conditions) | 38 | 15 | 0
Fever (General disorders and administration site conditions) | 5 | 2 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Flashing lights (Eye disorders) | 1 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0
Flu like symptoms (General disorders and administration site conditions) | 2 | 2 | 0
Fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Gait disturbance (General disorders and administration site conditions) | 0 | 1 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 4 | 3 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0
General disorders and administration site conditions - Other, specify (General disorders and administration site conditions) | 1 | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 7 | 11 | 0
Heart failure (Cardiac disorders) | 1 | 0 | 0
Hematoma (Vascular disorders) | 1 | 0 | 0
Hematuria (Renal and urinary disorders) | 2 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Hot flashes (Vascular disorders) | 2 | 2 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 10 | 10 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 6 | 5 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 3 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 3 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 7 | 6 | 0
Hypothyroidism (Endocrine disorders) | 3 | 5 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 2 | 0
Infusion related reaction (General disorders and administration site conditions) | 2 | 0 | 0
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 5 | 2 | 0
Intracranial hemorrhage (Nervous system disorders) | 1 | 0 | 0
Investigations - Other, specify (Investigations) | 0 | 1 | 0
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 2 | 0
Lipase increased (Investigations) | 0 | 1 | 0
Localized edema (General disorders and administration site conditions) | 1 | 1 | 0
Lung infection (Infections and infestations) | 2 | 3 | 0
Lymphedema (Vascular disorders) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 3 | 1 | 0
Mitral valve disease (Cardiac disorders) | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 2 | 2 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0
Nausea (Gastrointestinal disorders) | 13 | 11 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 2 | 0
Non-cardiac chest pain (General disorders and administration site conditions) | 2 | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0
Pain (General disorders and administration site conditions) | 4 | 7 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 5 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Papulopustular rash (Infections and infestations) | 2 | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 2 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 1 | 0
Personality change (Psychiatric disorders) | 1 | 0 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Platelet count decreased (Investigations) | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 11 | 0
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 5 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 | 7 | 0
Rash pustular (Infections and infestations) | 0 | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 | 3 | 0
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Retroperitoneal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 9 | 5 | 0
Skin infection (Infections and infestations) | 2 | 4 | 0
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 2 | 0
Thromboembolic event (Vascular disorders) | 1 | 3 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Tracheal fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 5 | 4 | 0
Urinary frequency (Renal and urinary disorders) | 2 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 3 | 0
Urinary tract pain (Renal and urinary disorders) | 2 | 0 | 0
Urinary urgency (Renal and urinary disorders) | 1 | 0 | 0
Uterine hemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal infection (Infections and infestations) | 1 | 0 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 1 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vasovagal reaction (Nervous system disorders) | 0 | 1 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 6 | 0
Weight gain (Investigations) | 5 | 1 | 0
Weight loss (Investigations) | 2 | 5 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/73/NCT03203473/Prot_SAP_000.pdf